CLINICAL TRIAL: NCT02233595
Title: Evaluation of Rectal Cancer Treatment Response Using PET/MRI
Acronym: Rectal PET/MRI
Status: Terminated | Type: Observational
Why Stopped: Low Accrual
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 144513; NCI-2015-00980 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2014-09-03; First posted 2014-09-08 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Rectal Adenocarcinoma
Keywords: MRI; PET; rectal cancer; adjuvant chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adjuvant chemotherapy
  Interventions: Radiation: Chemoradiation

INTERVENTIONS:
Radiation: Chemoradiation

SUMMARY:
The investigators will be using the combination of FDG-PET and multiparametric MRI in pre- and post-adjuvant chemoradiation therapy in order to attempt to predict pathologic response on surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of histopathologically confirmed rectal adenocarcinoma.
* Locally advanced disease as determined by ERUS or pelvic MRI. Endoscopy reports should clearly state both the T and N stage.
* Patients with cT2N1-3M0 or cT2-4NxM0 will be considered eligible for participation.
* Age ≥18.
* Ability to understand a written informed consent document and the willingness to sign it.
* Tumor must be determined to be surgically resectable. Surgical resection is planned to take place at Univeristy of California, San Francisco (UCSF).
* Neoadjuvant chemoradiation prior to resection is planned..
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.

Exclusion Criteria:

* ERUS tumor state of T1.
* Radiographic evidence of metastatic disease
* Weight in excess of limitations of the scanner or girth that prohibits entry into the bore of the PET/CT scanner due to size.
* Any medical condition which impairs the ability to lie flat and without movement for 15 minutes (e.g. cough, severe arthritis, etc.)
* Prior receipt of any therapy, including local excision, radiation or chemotherapy, for the diagnosed rectal adenocarcinoma.
* Prior history of pelvic radiation.
* Uncontrolled hyperglycemia (defined as inability to achieve a glucose of <250 mg/dL at time of fluorodeoxyglucose (FDG) injection).
* Impaired renal function (CKD 4 or 5: estimated glomerular filtration rate (eGFR) < 30 mLs/min), which is a contraindication to gadolinium containing contrast.
* Known allergy to gadolinium containing contrast agents.
* Contraindication to use of fluoropyrimidines as a radiosensitizing agent.
* Pregnancy or nursing. Women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to randomization. This is because of the potential teratogenic effects of the involved imaging modalities, radiation, and chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients with newly diagnosed rectal adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2018-01-28 (Actual)

PRIMARY OUTCOMES:
change in SUVmax | 2 months
  To determine whether percent change in SUVmax correlates with the extent of pathologic primary tumor response
tumor volume | 2 months
  To determine whether percent change in tumor volume correlates with the extent of pathologic primary tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Imaging Center at China Basin, San Francisco, California, United States